CLINICAL TRIAL: NCT06154057
Title: Retrospective Observational Study of Implant-supported Restorations With Implants Produced by Additive Manufacturing
Brief Title: Retrospective Observational Study of Implant-supported Restorations With Dental Implants.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M3 Health (Industry)
Collaborators: University of Guarulhos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Plenum Oss 002
Record Dates: First submitted 2023-11-14; First posted 2023-12-01 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-11

CONDITIONS: Oral Surgical Procedures
Keywords: Dental Implants; Synthetic Bone Graft; Additive Manufacture; Bone Loss; Success Rate
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dental Implants installed in an grafted area (sinus lifting) (Experimental): Dental implants produced by additive manufacturing installed in an area grafted with synthetic bone graft (Plenum® Osshp) - sinus lifting.
  Interventions: Procedure: Dental Implants installed in an grafted area (sinus lifting)
- Dental Implants installed in an grafted area (ridge augmentation) (Experimental): Dental implants produced by additive manufacturing installed in an area grafted with synthetic bone graft (Plenum® Osshp) - ridge augmentation.
  Interventions: Procedure: Dental Implants installed in an grafted area (ridge augmentation)
- Dental Implants installed in an grafted area (extraction sites) (Experimental): Dental implants produced by additive manufacturing installed in an area grafted with synthetic bone graft (Plenum® Osshp) - extraction sites (socket preservation or dental implant preparation/placement).
  Interventions: Procedure: Dental Implants installed in an grafted area (extraction sites)

INTERVENTIONS:
Procedure: Dental Implants installed in an grafted area (sinus lifting) — The patient will be invited to participate in the clinic to assess radiographic bone loss and clinical follow-up for 12 months.
  Other Names: maxillary sinus lift
  Arms: Dental Implants installed in an grafted area (sinus lifting)
Procedure: Dental Implants installed in an grafted area (ridge augmentation) — The patient will be invited to participate in the clinic to assess radiographic bone loss and clinical follow-up for 12 months.
  Other Names: Guided bone regeneration
  Arms: Dental Implants installed in an grafted area (ridge augmentation)
Procedure: Dental Implants installed in an grafted area (extraction sites) — The patient will be invited to participate in the clinic to assess radiographic bone loss and clinical follow-up for 12 months.
  Other Names: Guided bone regeneration
  Arms: Dental Implants installed in an grafted area (extraction sites)

SUMMARY:
This retrospective study aims to value the bone loss and the success and survival of the dental implants produced by additive manufacturing installed in an area grafted with Plenum® Osshp (synthetic bone graft). In addition, the biological and biomechanical performance of implant restorations supported through an observational retrospective solution will be observed. From 50 to 100 survey participants will be selected, who will be invited to attend the clinic for clinical, radiographic, and prosthetic evaluation and successful parameters between baseline, 3, 6, and 12 months. The data obtained regarding bone loss (primary outcome) of the analyzed regions and implant success and survival in area grafted with Plenum® Osshp (secondary outcome) will be evaluated by the paired t-test for the evaluation of the times (3, 6, and 12 months) and survival curves of the installed dental implants.

ELIGIBILITY:
Inclusion Criteria:

Clinical parameters:

* Presence or absence of pain or tenderness
* Presence or absence of suppuration or exudation
* Presence or absence of mobility

Prosthetic parameters

- Presence or absence of mechanical complications (problems in prefabricated components such as screws and abutments).

Radiographic Parameters

* Presence or absence of peri-implant radiolucidity.
* maintenance and quality of the bone graft volume in the grafted area to each clinical indication: ridge augmentation, extraction sites (socket preservation or dental implant preparation/placement) and sinus lifting.
* Distance between the shoulder of the implant and the first visible bone contact (in mm).
* Presence or absence of technical complications such as fracture or loss of porcelain structures.

Success Parameters

* Absence of pain or tenderness.
* Absence of suppuration or exudation.
* Clinical absence of implant mobility.
* Absence of peri-implant radiolucency.
* Minor loss of up to 1.5mm in the first year of function.
* Absence of mechanical or technical complications in the dental implant and in the prosthesis to the dental implants installed in an area grafted.

Exclusion Criteria:

* N/A

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The survival rate of dental implants produced by additive manufacturing installed in pristine bone and grafted areas with synthetic bone graft (Plenum® Osshp). | 12 months
  The main outcome is the survival rate (%) of successful implant-supported restoration after at least 1-year of occlusal loading (less than 0.5mm of bone loss)

SECONDARY OUTCOMES:
The survival rate of dental implants produced by additive manufacturing installed in different areas grafted with synthetic bone grafts (Plenum® Osshp) | 12 months
  Survival rate (%) of successful implant-supported restorations (less than 0.5mm of bone loss) placed in different bone areas (pristine bone, grafted areas with Plenum Oss including maxillary sinus augmentation, guided bone regeneration for both vertical and horizontal augmentation, and extraction sockets).
Rate of bone loss | 12 months
  A periapical x-ray will be performed at the implant placement region to check the bone level concerning the implant platform. Then, a vertical line will be drawn from the initial line to the bone level for measurement (mm). Standardized intraoral periapical radiographs will be obtained using a dental X-ray machine with a 35 cm long cone. The exposure parameter was 70 kV (Peak), 15mA, and 1/4s at a focus-sensor distance of 30cm. The X-rays will be captured with a digital camera and transferred to a personal computer. Image processing software will be used to store the scanned images. Subsequently, the images will be made available on a monitor and a linear measurement will be performed with software.

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Shibli, PhD, Principal Investigator — University of Guarulhos, UnG
Locations (1):
- University of Guarulhos, Guarulhos, São Paulo, Brazil